CLINICAL TRIAL: NCT01699984
Title: THE HOSPITALIZATION OF OLDER PATIENTS: RISK FACTORS, ADVERSE EVENTS AND OUTCOMES. A MULTICENTRE STUDY.
Brief Title: PERDOVE ANZIANI: a Prospective Cohort Study on Older Patients
Status: Completed | Type: Observational
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Responsible Party: Principal Investigator, Giovanni de Girolamo, M.D., M.D., Scientific Director, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Other Study IDs: 2012-1-PEV
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Dementia; Motor Impairments; Stroke; Thighbone Fractures
Keywords: Cognitive impairment.; Geriatrics.; Hospital admission.; Hospital discharge.
MeSH Terms: conditions — Dementia; Stroke; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for the assessment of APOE genetic polymorphisms; routine lab examinations.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hospitalized patients: All patients hospitalized in 4 inpatient facilities in Northern Italy during 4 index-months.

SUMMARY:
This prospective observational cohort study aims at studying functional and clinical outcomes of patients (N = 329) admitted to 4 geriatric hospital facilities of the St John of God Order in Northern Italy during an index period of 4 months. Other areas assessed include variables that help or hinder the discharge of patients with sufficient residential autonomy and the predictive ability of clinicians compared with the evaluation of selective indicators of outcome (clinical and instrumental).

Patients are followed from the first day of hospitalization until discharge or up to 3 months and 1 day after the date of admission ("long-term care" patients).

At admission a "Patient Form" including social, demographic and clinical informations and a series of standardized assessment tools is completed with the help of clinicians, nurses and caregivers (when available).

For each patient, during hospitalization, an analysis of apolipoprotein ApoE polymorphisms is performed and adverse events occurred during hospitalization are monitored, as well as the predictive abilities of clinicians and any recent CT and MRI. Patients are reassessed at discharge (or after 3 months for "long-term care" patients) and at 6 months follow-up of with a standardized telephone interview to assess clinical and functional status and possible changes in the residential status of the patient.

ELIGIBILITY:
Inclusion Criteria:

* age 65 or older
* informed consent provided

Exclusion Criteria:

* younger than 65 years
* informed consent not provided

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 or older admitted to 4 geriatric inpatient facilities.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
evaluation of clinical improvement | from admission to discharge (or after 3 months of hospitalization) and 6 months follow-up

SECONDARY OUTCOMES:
identification of variables predictive of outcomes | at discharge (or 3 months after admission) and 6 months follow-up

OTHER OUTCOMES:
evaluation of predictive abilities of clinicians | admission, discharge (or 3 months of hospitalization) and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni de Girolamo, M.D., Principal Investigator — IRCCS Centro San Giovanni di Dio Fatebenefratelli
Locations (4):
- Italy (4):
  - IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Brescia
  - Sacro Cuore di Gesù Centre, San Colombano al Lambro, Milan
  - beata Vergine della Consolata Hospital, San Maurizio Canavese, Turin
  - San Raffaele Arcangelo Hospital, Venezia, Venezia

REFERENCES:
- See also: Website of the coordinating centre — http://www.irccs-fatebenefratelli.it